CLINICAL TRIAL: NCT03119805
Title: Defining Cut-off Values for Widely-used Composite Scores and Patient-reported Outcome Measures in Psoriatic Arthritis Corresponding to Remission and Flare Assessed by the Physician and the Patient
Brief Title: Remission and Flare in Psoriatic Arthritis: a Prospective 6-month Study With a Double Perspective.
Acronym: ReFlaP
Status: Completed | Type: Observational
Sponsor: Groupe Hospitalier Pitie-Salpetriere (Other)
Responsible Party: Principal Investigator, Laure Gossec, Professor, Groupe Hospitalier Pitie-Salpetriere
Other Study IDs: ongoing
Record Dates: First submitted 2017-01-04; First posted 2017-04-19 (Actual); Last update posted 2018-10-17 (Actual); Status verified 2018-10

CONDITIONS: Psoriatic Arthritis
Keywords: composite scores; patient reported outcomes; patient perpective; physician perspective; cut-off values; flare; remission; minimal disease activity; low disease activity
MeSH Terms: conditions — Arthritis, Psoriatic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study is to define cut-off values of the most widely used composite scores and patient-reported outcomes, for levels corresponding to remission/low disease activity and for changes in levels corresponding to flares, in PsA, when remission/low disease activity and flare are defined from the patient and physician perspective. The ReFlaP (Remission/Flare in PsA) study is a prospective, multicentric international, longitudinal, observational study.

DETAILED DESCRIPTION:
Introduction: Psoriatic arthritis (PsA) is a heterogeneous chronic disease with a significant patient-perceived impact leading to pain, fatigue, impaired function and quality of life and psychological distress. Remission is the announced treatment target in PsA. Several definitions of remission have been proposed including definitions on composite scores such as the Disease Activity in Psoriatic Arthritis (DAPSA) and Minimal Disease Activity (MDA), however their translation into the patient's perspective is lacking. Flares are frequent in PsA and are important for patients but are not well-defined from the physician's perspective. Although some work is ongoing regarding remission and flare from the patient's perspective, currently no information allows to cross-tabulate and compare the patient and physician perspectives regarding remission and flare in PsA .

The objective is to define cutoffs of the most widely used composite scores and PROs, for levels corresponding to remission/low disease activity and for changes in levels corresponding to flares, in PsA, when remission/low disease activity and flare are defined from the patient and physician perspective.

Methods Design: the ReFlaP (Remission/Flare in PsA) study is a prospective, multicentric international, longitudinal, observational study. It will take place in 2017-18 in 25 centers across Europe, North and South America and Asia. Investigators plan to include a total of 450 patients. The inclusion period will last 6 months; each center will include around 20 patients. Each patient is seen twice at baseline and at 1-6 months (follow-up visit) in the context of usual care.

Patients: Consecutive adult patients with definite PsA (according to ClASsification of Psoriatic ARthritis (CASPAR) criteria and confirmation by a rheumatologist), more than 2 years of disease duration, and will be included after signed informed consent.

Data collection: During each visit, physicians will collect data on the disease and on disease activity: 66 swollen joint counts, 68 tender joint counts, tender entheseal points (Leeds Enthesitis Index) and body surface area of psoriasis. This will allow calculation of most of the usual composite scores of PsA: Arythmetic Mean of Desirability Functions modified (AMDF modified), Disease Activity in PSoriatic Arthritis (DAPSA), clinical DAPSA (c-DAPSA), Minimal Disease Activity (MDA) and Psoriatic Arthritis Disease Activity Score (PASDAS). Well-validated Patient Reported Outcomes will be collected from patients: Patient Global Assessment (PGA), Pain, Health Assessment Quality (HAQ), PSoriatic Arthritis Impact of Disease (PSAID), Psoriatic Arthritis Quality of Life (PsAQoL), 12-Item Short Form Health Survey (SF-12), Patient Acceptable Symptom State (PASS) and Minimal clinically important differences (MCID) as well as the recent Flare questionnaire proposed by GRAPPA. Assessment of disease activity status (i.e. remission or flare) will be performed by both physician and patient using global questions.

Planned analysis

To define cutoffs of the most widely used composite scores and PROs, for levels corresponding to remission/low disease activity and for changes in levels corresponding to flares, in PsA:

From the health professional perspective, the gold standard for 'remission' will be MDA and sensitivity analyses will use physician-perceived remission/low disease activity (single questions) and remission in composite scores (DAPSA, c-DAPSA, modified AMDF, PASDAS); for flare the gold standard will be decision of treatment intensification and sensitivity analyses will use: global assessment of flare and increase in category of disease activity in the composite scores.

From the perspective of the patient, the gold standard will be for 'remission', PASS and as sensitivity analysis, patient-perceived remission/low disease single questions yes/no, and for flares, the GRAPPA flare questionnaire, and as sensitivity analyses, flare according to the patient (single question) and the assessment of worsening in MCID.

Investigators will assess what physician-defined remission/low disease activity/flare and patient-defined remission/low disease activity/flare correspond to both on composite 'physician' scores and on all the collected PRO scores. Investigators will use data collected at baseline cross sectionally for remission/low disease activity and changes in scores between the 2 visits for flares.

Cutoff values for each outcome and for each change in outcome will be calculated using ROC curves and 75th percentile analyses. Sensitivity analyses will explore cutoff values found according to patient demographic characteristics and country. Investigators will compare attainment of remission or flare according to the different definitions, using kappa analyses. Rasch analyses will be used as necessary.

Planned outcomes The expected outcomes of this study are a better knowledge of remission/low disease activity and flare in PsA in accordance to the perspectives of patients and physicians. Investigators will define cutoff values for most widely-used scores in PsA, allowing easier interpretation of study results and in the clinic, helping a better communication with patients.

Better knowledge of the important aspects of disease fluctuation and of patient relevant disease targets in PsA should enhance patient care and management in a treat-to-target approach.

ELIGIBILITY:
Inclusion Criteria:

* Age>18 years
* Definite PsA according to the ClASsification of Psoriatic ARthritis (CASPAR) criteria and diagnosis confirmed by a rheumatologist. (Taylor2006)
* Willingness to participate and signed informed consent.
* There are no inclusion criteria based on disease activity or treatment
* Patients with more than 2 years of disease duration will be included in the study for more homogeneity.

Patient will be included consecutively. A registry will be kept locally to note the age and gender of patients who have been proposed the study but refused to participate.

Exclusion Criteria:

* No definite PsA or less than 2 years of disease duration
* Patients who don't speak or read the local language or are not comfortable filling in a paper CRF in the local language.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Over the 6 months recruitment period, all patients with definite PsA who satisfy the inclusion criteria, seen in outpatient visits in the participating centers by one of the investigators, will be asked to participate. It is planned to take place in 6 participating centres in France, 15 other European tertiary rheumatology centers (Germany, Hungary, Ireland, Italy, Norway, Romania, Spain, Turkey and the UK), 4 centers in the USA, 2 centers in Canada, 1 in Brazil, and 2 in Asia (Singapore and Russia).It is planned that in each center, 15-30 patients will be included. The first 15-30 consecutive patients will be selected in each center to reduce bias selection.
Sampling Method: Probability Sample
Enrollment: 466 (Actual)
Dates: Start 2017-05-18 (Actual); Primary Completion 2018-01-30 (Actual); Study Completion 2018-07-30 (Actual)

PRIMARY OUTCOMES:
To determine the cutoff value of PsAID corresponding to flare | 6 months
  For flare, the gold standard will be decision of treatment intensification. The primary outcome will be to determine the cutoff value of PsAID corresponding flare.
  The PsAID is a questionnaire (paper CRF) that can be used to calculate a score reflecting the impact of psoriatic arthritis (PsA) from the patients' perspective. (Gossec L et al., A patient-derived and patient-reported outcome measure for assessing psoriatic arthritis: elaboration and preliminary validation of the Psoriatic Arthritis Impact of Disease (PsAID) questionnaire, a 13-country EULAR initiative. Ann Rheum Dis. 2014;73(6):1012-9).
To determine the cutoff value of PsAID corresponding to remission | 6 months
  For remission, the gold standard will be Minimal Disease Activity. The primary outcome will be to determine the cutoff value of PsAID corresponding to remission. Patients are classified as achieving Minimal Disease Activity if they fulfill 5 of 7 outcome measures: tender joint count ≤1; swollen joint count ≤1; psoriasis activity and severity index ≤1 or body surface area ≤3; patient pain visual analog scale (VAS) score of ≤15; patient global disease activity VAS score of ≤20; Health Assessment Questionnaire (HAQ) score ≤0.5; and tender entheseal points ≤1. (L C Coates, J Fransen, P S Helliwell Defining minimal disease activity in psoriatic arthritis: a proposed objective target for treatment Clinical and epidemiological research Ann Rheum Dis 2010;69:48-53.)

CONTACTS AND LOCATIONS:
Locations (22):
- United States (2):
  - Ana- Maria Orbai, Baltimore, Maryland
  - Husni, Cleveland, Ohio
- Smolen, Vienna, Austria
- Palominos, Porto Alegre, Brazil
- Canada (3):
  - Aydin, Ottawa
  - Sibel Aydin, Ottawa
  - Eder, Toronto
- Talli, Tallinn, Estonia
- France (5):
  - Soubrier, Clermont-Ferrand
  - Dernis, Le Mans
  - Laure Gossec, Paris
  - Richette, Paris
  - Ruyssen-Witrand, Toulouse
- Uta Kiltz, Herne, Germany
- Italy (2):
  - Lubrano, Campobasso
  - Rossana Scrivo, Roma
- Balanescu, Bucharest, Romania
- Inna Gaydukova, Saratov, Russia
- Katy Leung, Singapore, Singapore
- Juan Canete, Barcelona, Spain
- Kalyoncu, Ankara, Turkey (Türkiye)
- Laura Coates, Oxford, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yazji SM, Helliwell PS, Balanescu A, Dernis E, Kiltz U, Kalyoncu U, Leung YY, Orbai AM, Smolen JS, de Wit M, Gossec L, Coates LC. Association Between Patient Perception of Disease Status and Different Components of the Minimal Disease Activity Criteria in Psoriatic Arthritis. J Rheumatol. 2025 Apr 1;52(4):362-367. doi: 10.3899/jrheum.2024-1149. PMID 39814446
- [Derived] Leung YY, Eder L, Orbai AM, Coates LC, de Wit M, Smolen JS, Kiltz U, Palominos P, Canete JD, Scrivo R, Balanescu A, Dernis E, Meisalu S, Soubrier M, Kalyoncu U, Gossec L. Association between obesity and likelihood of remission or low disease activity status in psoriatic arthritis applying index-based and patient-based definitions of remission: a cross-sectional study. RMD Open. 2023 Sep;9(3):e003157. doi: 10.1136/rmdopen-2023-003157. PMID 37709527
- [Derived] Lucasson F, Kiltz U, Kalyoncu U, Leung YY, Palominos P, Canete JD, Scrivo R, Balanescu A, Dernis E, Meisalu S, Ryussen-Witrand A, Soubrier M, Aydin SZ, Eder L, Gaydukova I, Lubrano E, Richette P, Husni E, Coates LC, de Wit M, Smolen JS, Orbai AM, Gossec L. Disparities in healthcare in psoriatic arthritis: an analysis of 439 patients from 13 countries. RMD Open. 2022 May;8(1):e002031. doi: 10.1136/rmdopen-2021-002031. PMID 35523519
- [Derived] Coates LC, Robinson DE, Orbai AM, Kiltz U, Leung YY, Palominos P, Canete JD, Scrivo R, Balanescu A, Dernis E, Meisalu S, Ruyssen-Witrand A, Eder L, de Wit M, Smolen JS, Lubrano E, Gossec L. What influences patients' opinion of remission and low disease activity in psoriatic arthritis? Principal component analysis of an international study. Rheumatology (Oxford). 2021 Nov 3;60(11):5292-5299. doi: 10.1093/rheumatology/keab220. PMID 33751029
- [Derived] Orbai AM, Perin J, Gorlier C, Coates LC, Kiltz U, Leung YY, Palominos PE, Canete JD, Scrivo R, Balanescu A, Dernis E, Talli S, Ruyssen-Witrand A, Soubrier M, Aydin S, Eder L, Gaydukova I, Lubrano E, Kalyoncu U, Richette P, Husni ME, Smolen JS, de Wit M, Gossec L. Determinants of Patient-Reported Psoriatic Arthritis Impact of Disease: An Analysis of the Association With Sex in 458 Patients From Fourteen Countries. Arthritis Care Res (Hoboken). 2020 Dec;72(12):1772-1779. doi: 10.1002/acr.24090. PMID 31609525
- [Derived] Gorlier C, Orbai AM, Puyraimond-Zemmour D, Coates LC, Kiltz U, Leung YY, Palominos P, Canete JD, Scrivo R, Balanescu A, Dernis E, Talli S, Ruyssen-Witrand A, Soubrier M, Aydin SZ, Eder L, Gaydukova I, Lubrano E, Kalyoncu U, Richette P, Husni ME, de Wit M, Smolen JS, Gossec L. Comparing patient-perceived and physician-perceived remission and low disease activity in psoriatic arthritis: an analysis of 410 patients from 14 countries. Ann Rheum Dis. 2019 Feb;78(2):201-208. doi: 10.1136/annrheumdis-2018-214140. Epub 2018 Nov 15. PMID 30442648

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-04-21): https://cdn.clinicaltrials.gov/large-docs/05/NCT03119805/Prot_SAP_000.pdf